CLINICAL TRIAL: NCT00660231
Title: A Phase II Study of Gemcitabine and Bexarotene (Gembex) in the Treatment of Cutaneous T-cell Lymphoma
Brief Title: Gemcitabine and Bexarotene in Treating Patients With Progressive or Refractory Stage IB, Stage II, Stage III, or Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma
Acronym: GemBex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/06/009; CRUK-UCL-GEMBEX; EU-20841; EUDRACT 2006-000591-33
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage IB mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage IB cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Bexarotene; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GemBex (Experimental): Gemcitabine days 1 and 8 of a 3 week cycle (4 cycles total - 12 weeks) Bexarotene daily: in combination with Gemcitabine during first 12 weeks, then Bexarotene maintenance until disease progression.
  Interventions: Drug: bexarotene; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: bexarotene — Bexarotene daily p.o. 150mg/sq m during week 1 and 2, then 300mg/sq m if tolerated.
  Other Names: Targretin
Drug: gemcitabine hydrochloride — Gemcitabine i.v. 1000mg/sq m day 1 and day 8 of four 21 day cycles.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and bexarotene, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying giving gemcitabine together with bexarotene to see how well it works in treating patients with progressive or refractory stage IB, stage II, stage III, or stage IV cutaneous T-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Confirm the feasibility and efficacy of the combination of gemcitabine hydrochloride and bexarotene in patients with cutaneous T-cell lymphoma whose disease is no longer controlled by skin-directed therapy and who have had at least one prior systemic therapy.

Secondary

* Determine the rate of objective disease control as defined by complete response (CR), clinical complete response (CCR), partial response (PR), and stable disease (SD) for 6 months as determined by the Objective Primary Disease Response Evaluation Criteria (OPDREC).
* Evaluate the duration and durability of objective disease response (CR, CCR and PR) as determined by OPDREC criteria.
* Evaluate time to objective disease response.
* Determine the safety of this combination in terms of adverse events, clinical laboratory data, physical examinations, rate of neutropenic fever and sepsis, blood transfusions, and treatment compliance.
* Determine the time to objective disease progression.
* Determine the time to treatment failure.
* Determine change from baseline in Severity-Weighted Assessment Tool (SWAT) value, Erythroderma SWAT value, Pruritus Visual Analogue Scale, and ECOG performance status.
* Determine proportion of disease control, response, and progression as determined by RECIST criteria.
* Evaluate the proportion of patients with clearing of Sézary cells from the blood and bone marrow.
* Measure changes in patient assessed Quality of Life using Skindex 29 and EORTC QLQ-30.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV on days 1 and 8 and oral bexarotene daily on days 1-21. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. After 4 courses of study therapy, patients with responding disease receive oral bexarotene alone daily until disease progression or treatment no longer tolerated.

Patients complete a quality of life questionnaire at baseline, during study therapy, and after completion of study treatment.

After completion of study treatment, patients are followed every 2 months for up to 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma (CTCL) including its variants (e.g., mycosis fungoides and Sézary syndrome)

  * CTCL stage IB, IIA, IIB, III or IVA disease
  * No visceral involvement (i.e., stage IVB disease)

    * Lymphadenopathy is allowed
* Patients must have developed progressive disease after receiving or have been refractory to at least 1 course of prior standard, systemic, skin-directed therapy (e.g., interferon, chemotherapy, or denileukin diftitox [Ontak®])
* No CD30 + (Ki1+ve) anaplastic large cell lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 6 months
* Hemoglobin ≥ 9.0 g/dL (transfusions and/or erythropoietin are allowed)
* ANC > 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 2 times ULN
* Serum creatinine ≤ 2 times ULN
* No clinically significant active infection
* No uncontrolled diabetes mellitus
* No excessive alcohol consumption
* No biliary tract disease
* No history of pancreatitis
* HIV negative
* Hepatitis B and C negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study participation
* No other malignancy within the past 5 years except curatively treated basal or squamous cell skin cancer, cervical epithelial neoplasm CIN1, or carcinoma in situ
* No other significant medical or psychiatric condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since any prior investigational agent
* More than 2 weeks since prior topical steroids or more than 4 weeks since prior systemic steroids
* Local radiotherapy may be given to isolated symptomatic tumour nodules that require immediate treatment for up to 2 weeks prior to study drugs
* No prior treatment with bexarotene (Targretin®)
* No concurrent anticancer therapy
* No concurrent investigational agent
* No concurrent drug therapy with other medications that can elevate triglycerides or cause pancreatic toxicity (e.g., gemfibrozil)
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Rate of objective response | at 24 weeks

SECONDARY OUTCOMES:
Duration and durability of objective disease response | up to 5 years after treatment start
  Time from first date of treatment to the first date of diagnosis of progressive disease
Assessment of quality of life | up to 5 years after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Tim Illidge, Principal Investigator — The Christie NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - St. Thomas' Hospital, London, England
  - Christie Hospital, Manchester, England
  - Southampton General Hospital, Southampton, England
  - Royal Cornwall Hospital, Truro, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland